CLINICAL TRIAL: NCT01314235
Title: The Influence of Clonidine on the Thrombozytes of Patients Under Double Anticagulation With ASS and Clopidogrel - an in Vitro Study
Brief Title: Influence of Clonidine on Thrombozytes of Blood of Patients Under Anticoagulation Therapy With ASS and Clopidogrel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Goethe University (Other)
Responsible Party: Philipp Schmidt, Goethe University
Other Study IDs: Clonidinstudy
Record Dates: First submitted 2011-03-08; First posted 2011-03-14 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Anticoagulation
Keywords: anticoagulation with ASS; anticoagulation with clopidogrel

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Clonidin works as a presynaptic agonist of alpha-sympathomimetic receptors of the brain but also in many other tissues. It is part of balanced anesthesia in general anesthesiology as well as a sedastive agent in intensive care units, but also serves as a third-line agent in many psychiatric diseases including ADHD, schizophrenia and PTSD.

The investigators want to show whether clonidin has an procoagulatoric effect on thrombozytes of patients under double anticoagulaotirc treatment with ASS and clopidogrel. The investigators will use a flowcytometric assay to determine activation of thrombozytes when they come into contact with clonidine in vitro as well as Multiplate analyses to determine activation of thrombozytes, either thrombin.induced aggregation, ADP-induced aggregation or arachidonic acid-induced aggregation of thrombozytes.

ELIGIBILITY:
Inclusion Criteria:

* Elective vascular surgical patients with long-term medication (at least 5 days) with ASS and clopidogrel
* Age above 18 years

Exclusion Criteria:

* Additional anticoagulatoric treatment woth another inhibitor of platelet aggregation
* Surgery within the last two weeks
* Patients with long-term mediaction with omeprazole
* Patients under hemodialysis
* Patients with renal insufficiency (creatinine above 1.5mg/dl, urea above 80mg/dl)
* Patients with hepatic dysfunction (GOT above 30U/I, GPT above 30 U/I, GLDH above 10 U/I)
* Age under 18 yeary
* Non-responder to ASS and / or clopidogrel

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients going under vascular surgery with anticagulation with both ASS and clopidogrel
Sampling Method: Non-Probability Sample
Dates: Start 2010-10

PRIMARY OUTCOMES:
Numbers of participants with an activated area under the curve in ASPI test | 30 minutes
  Blood of patients under ASS and clopidogrel will show an activated platelet aggregation due to titrated clonidine in ASPI test, i.e. an activated area under the curve in Multiplate analysis.

SECONDARY OUTCOMES:
Numbers of participants with an activated area under the curve in TRAP test and ADP test | 30 minutes
  Blood of patients under ASS and clopidogrel will show an activated platelet aggregation due to titrated clonidine in TRAP test and ADP test, i.e. an activated area under the curve in Multiplate analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Johann-Wolfgang-Goethe University, Frankfurt am Main, Hesse, Germany